CLINICAL TRIAL: NCT05325658
Title: Influence of Modified Diet, Exercise and Electrical Swallowing Muscle Stimulation on Swallowing Function and Quality of Life in Elderly Patients With Oropharyngeal Dysphagia
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Margarita Rugaitiene, Principal Investigator, Lithuanian University of Health Sciences
Other Study IDs: 2.3
Record Dates: First submitted 2021-09-29; First posted 2022-04-13 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Oropharyngeal Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Fees and Charges; Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oropharyngeal dysphagia: Patients with oropharyngeal dysphagia. Patients will be examined before and after combination therapy.
  Interventions: Other: FEES, treatment with modified diet, electrical swallowing muscle stimulation.

INTERVENTIONS:
Other: FEES, treatment with modified diet, electrical swallowing muscle stimulation. — Endoscopic swallowing assessment (FEES) consists of three parts:1) assessment of mouth, throat anatomy and more; 2) the patient is given to swallow a certain amount and consistency of liquids and solid food. 3) evaluated: preparation of the bolus for swallowing, aspiration. An 8-point Penetration-Aspiration scale is described.Swallowing exercises. Swallowing exercises are also used in practice, which can help coordinate the swallowing muscles or stimulate the nerves involved in the swallowing reflex.Transcutaneous electrical stimulation is a method of treating dysphagia in which weak electrical impulses stimulate the muscles in the neck area associated with swallowing. In patients with oropharyngeal dysphagia, patients have great difficulty swallowing water of normal consistency or other non-thick liquids, so they should be thickened with special thickeners to such an extent that the patient does not experience discomfort and be able to swallow.

SUMMARY:
Tasks of biomedical research:

1. To determine the severity of oropharyngeal dysphagia and the risk of aspiration in elderly patients.
2. To evaluate the quality of life of older patients with oropharyngeal dysphagia by performing validation of the Lithuanian version of the quality of life questionnaires in patients with oropharyngeal dysphagia.
3. To evaluate the severity of oropharyngeal dysphagia in elderly patients, the risk of aspiration, and quality of life after interventions.

Data on the sex, age and disease of the swallowing disorder will be collected. No processing of other personal data and health indicators is planned. All data will be collected in questionnaires. The data will be depersonalized by giving the patient a code.

The results and conclusions of the research will be described in the doctoral dissertation and will be used for scientific articles.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years of age and older;
* Swallowing disorder suspected during hospitalization - oropharyngeal dysphagia;
* Patient's written consent.

Exclusion Criteria:

* severe oropharyngeal dysphagia (when feeding into the stomach through a nasogastric tube is required);
* Significant respiratory or heart failure: dyspnoea (respiratory rate> 20 rpm, SpO2 <90%), tachycardia (HR> 100 rpm);
* very severe malnutrition (severe exhaustion, severe signs of sarcopenia);
* final stage of oncological disease;
* severe dementia (Short Mental Test (MMSE) <10 points);
* Ingestion assessment with a fibroendoscope (FEES) did not reveal any swallowing problems (no dysphagia).

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Geriatric patients treated at Kaunas Hospital who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the influence of modified diet, exercise and electrical swallowing muscle stimulation on swallowing function and quality of life in elderly patients with oropharyngeal dysphagia. | 2021-2024
  Primary outcomes focus on domains within reduction in the severity of oropharyngeal dysphagia and a reduction in the risk of aspiration after administration of a modified diet, electrical swallowing muscle stimulation and exercise to improve swallowing, after 10 days. The Penetration - Aspiration (J.C. Rosenbek et al., 1996) scale will be used before and after treatment to evaluate FEES. Assessing FEES: The higher the score, the more severe the disease.
Evaluation of the influence of modified diet, exercise and electrical swallowing muscle | 2021-2024
  Dysphagia Handicap Index (DHI): The higher the score, the more severe oropharyngeal dysphagia.
Evaluation of the influence of modified diet, exercise and electrical swallowing muscle | 2021-2024
  SWAL-QoL / SWAL-CARE: frequency scale (in questions 3, 5, 6, 9) and an evaluation scale (in questions 1, 2, 4, 7, 8), in the form of a 5-point Likert scale, where 1 corresponds to worst QoL and 5 to best QoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Margarita Rugaitienė, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided